CLINICAL TRIAL: NCT03620162
Title: A Phase 3, Multicenter, Randomized, Double-blind Study to Evaluate the Interchangeability of V114 and Prevnar 13™ With Respect to Safety, Tolerability, and Immunogenicity in Healthy Infants (PNEU-DIRECTION)
Brief Title: A Study to Evaluate the Interchangeability of V114 and Prevnar 13™ in Healthy Infants (V114-027/PNEU-DIRECTION)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-027; V114-027 (Other: Merck); 2018-001151-12 (EudraCT Number)
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Results first posted 2021-08-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine; RotaTeq; Rotavirus Vaccines; pentacel; Recombivax HB; Hepatitis B Vaccines; Hiberix; Chickenpox Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL intramuscular (IM) injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants will concomitantly receive other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
  Interventions: Biological: Prevnar 13™; Biological: RotaTeq™; Biological: Pentacel™; Biological: RECOMBIVAX HB™; Biological: HIBERIX™; Biological: M-M-R™ II; Biological: VARIVAX™
- Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 (Experimental): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and a single 0.5 mL IM injection of V114 on Months 10-13 (Vaccination 4). Participants will concomitantly receive other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
  Interventions: Biological: Prevnar 13™; Biological: V114; Biological: RotaTeq™; Biological: Pentacel™; Biological: RECOMBIVAX HB™; Biological: HIBERIX™; Biological: M-M-R™ II; Biological: VARIVAX™
- Group 3: Prevnar 13™-Prevnar 13™-V114-V114 (Experimental): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2) and a single 0.5 mL IM injection of V114 on Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants will concomitantly receive other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
  Interventions: Biological: Prevnar 13™; Biological: V114; Biological: RotaTeq™; Biological: Pentacel™; Biological: RECOMBIVAX HB™; Biological: HIBERIX™; Biological: M-M-R™ II; Biological: VARIVAX™
- Group 4: Prevnar 13™-V114-V114-V114 (Experimental): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of V114 on Month 2 (Vaccination 2), Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants will concomitantly receive other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
  Interventions: Biological: Prevnar 13™; Biological: V114; Biological: RotaTeq™; Biological: Pentacel™; Biological: RECOMBIVAX HB™; Biological: HIBERIX™; Biological: M-M-R™ II; Biological: VARIVAX™
- Group 5: V114-V114-V114-V114 (Experimental): Participants will receive a single 0.5 mL IM injection of V114 on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants will concomitantly receive other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
  Interventions: Biological: V114; Biological: RotaTeq™; Biological: Pentacel™; Biological: RECOMBIVAX HB™; Biological: HIBERIX™; Biological: M-M-R™ II; Biological: VARIVAX™

INTERVENTIONS:
Biological: Prevnar 13™ — Prevnar 13™ contains the pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg each) and 6B (4.4 mcg) in each 0.5 mL dose given via IM injection.
  Arms: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™; Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Group 4: Prevnar 13™-V114-V114-V114
Biological: V114 — V114 contains the pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (2 mcg each), and serotype 6B (4 mcg) in each 0.5 mL dose given via IM injection.
  Other Names: VAXNEUVANCE™
  Arms: Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Group 4: Prevnar 13™-V114-V114-V114; Group 5: V114-V114-V114-V114
Biological: RotaTeq™ — RotaTeq™ live, pentavalent Rotavirus vaccine given as background treatment via oral solution.
  Other Names: V260; trade names of the concomitant vaccines may vary depending on where clinical supplies are sourced.
Biological: Pentacel™ — Pentacel™ Diphtheria and Tetanus Toxoids and Acellular Pertussis Adsorbed, Inactivated Poliovirus and Haemophilus b Conjugate (Tetanus Toxoid Conjugate) Vaccine, given as background treatment via IM injection in the opposite limb to V114 and Prevnar 13™ administration.
  Other Names: Trade names of the concomitant vaccines may vary depending on where clinical supplies are sourced.
Biological: RECOMBIVAX HB™ — RECOMBIVAX HB™ Hepatitis B Vaccine (Recombinant), given as background treatment via IM injection in the opposite limb to V114 and Prevnar 13™ administration.
  Other Names: V232, HEPTAVAX™-II, HBVAXPRO; trade names of the concomitant vaccines may vary depending on where clinical supplies are sourced.
Biological: HIBERIX™ — HIBERIX™ Haemophilus b Conjugate Vaccine (Tetanus Toxoid Conjugate), given as background treatment via IM injection in the opposite limb to V114 and Prevnar 13™ administration.
  Other Names: Trade names of the concomitant vaccines may vary depending on where clinical supplies are sourced.
Biological: M-M-R™ II — M-M-R™ II (Measles, Mumps, and Rubella Virus Vaccine Live), given as background treatment via subcutaneous (SC) injection in the opposite limb to V114 and Prevnar 13™ administration.
  Other Names: V205C; trade names of the concomitant vaccines may vary depending on where clinical supplies are sourced.
Biological: VARIVAX™ — VARIVAX™ Varicella Virus Vaccine Live, given as background treatment via SC injection in the opposite limb to V114 and Prevnar 13™ administration.
  Other Names: V210; trade names of the concomitant vaccines may vary depending on where clinical supplies are sourced.

SUMMARY:
The goal of this study is to evaluate the safety, tolerability, and immunogenicity of the Pneumococcal Conjugate Vaccines (PCVs) V114 and Prevnar 13™ in healthy infants switched from Prevnar 13™ to V114 during the four-dose PCV immunization schedule.

ELIGIBILITY:
Inclusion Criteria:

* Is Healthy, based on clinical judgment of the investigator
* Has a legally acceptable representative who understands the study procedures, alternate treatments available, and risks involved with the study and voluntarily agrees to participate by giving written informed consent.

Exclusion Criteria:

* Has a history of invasive pneumococcal disease (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease
* Has a known hypersensitivity to any component of the pneumococcal conjugate vaccine (PCV), any component of the licensed pediatric vaccines to be administered concomitantly in the study, or any diphtheria toxoid-containing vaccine
* Has any contraindication to the concomitant study vaccines being administered in the study
* Has a known or suspected impairment of immunological function
* Has a history of congenital or acquired immunodeficiency
* Has or his/her mother has a documented human immunodeficiency virus (HIV) infection
* Has or his/her mother has a documented hepatitis B surface antigen - positive test
* Has known or history of functional or anatomic asplenia
* Has failure to thrive based on the clinical judgment of the investigator
* Has a known coagulation disorder contraindicating intramuscular vaccination
* Has a history of autoimmune disease (including but not limited to systemic lupus erythematosus, antiphospholipid syndrome, Behcet's disease, autoimmune thyroid disease, polymyositis and dermatomyositis, scleroderma, type 1 diabetes mellitus, or other autoimmune disorders)
* Has a known neurologic or cognitive behavioral disorder, including encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive development disorder, and related disorders
* Has received a dose of any pneumococcal vaccine prior to study entry
* Has received >1 dose of monovalent hepatitis B vaccine or hepatitis B based combination vaccine prior to study entry
* Has received a dose of rotavirus vaccine prior to study entry
* Has received a blood transfusion or blood products, including immunoglobulins
* Has participated in another clinical study of an investigational product before the beginning or anytime during the duration of the current clinical study
* Has any other reason that, in the opinion of the investigator, may interfere with the evaluation required by the study
* Has an immediate family member (e.g., parent/legal guardian or sibling) who is investigational site or Sponsor staff directly involved with this study.

Ages: 42 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 900 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (34):
- United States (22):
  - Alabama Clinical Therapeutics ( Site 0015), Birmingham, Alabama
  - Southeastern Pediatric Associates, P.A. ( Site 0002), Dothan, Alabama
  - Children's Clinic of Jonesboro, PA ( Site 0022), Jonesboro, Arkansas
  - Davita Medical Group ( Site 0012), Colorado Springs, Colorado
  - Suncoast Research Associates, LLC ( Site 0035), Miami, Florida
  - Kentucky Pediatric/Adult Research Inc ( Site 0011), Bardstown, Kentucky
  - Pediatric Associates of Fall River ( Site 0021), Fall River, Massachusetts
  - Midwest Children's Health Research Institute, LLC ( Site 0024), Lincoln, Nebraska
  - Midwest Children's Health Research Institute, LLC ( Site 0003), Lincoln, Nebraska
  - Midwest Children's Health Research Institute, LLC ( Site 0004), Lincoln, Nebraska
  - Midwest Children's Health Research Institute, LLC ( Site 0001), Lincoln, Nebraska
  - Summerwood Pediatrics ( Site 0009), Liverpool, New York
  - University of Rochester Medical Center ( Site 0029), Rochester, New York
  - SUNY Upstate Medical University ( Site 0008), Syracuse, New York
  - Piedmont Healthcare, PA ( Site 0025), Statesville, North Carolina
  - Coastal Pediatric Research ( Site 0006), Charleston, South Carolina
  - Parkside Pediatric ( Site 0007), Greenville, South Carolina
  - Holston Medical Group ( Site 0018), Kingsport, Tennessee
  - Ventavia Research Group LLC ( Site 0017), Fort Worth, Texas
  - University of Texas Medical Branch ( Site 0023), Galveston, Texas
  - Wasatch Pediatrics-Cottonwood Office ( Site 0014), Murray, Utah
  - Multicare ( Site 0019), Spokane, Washington
- Puerto Rico (5):
  - Cooperativa de Facultad Medica Sanacoop ( Site 0057), Bayamón
  - Clinical Research of Puerto Rico ( Site 0050), Guayama
  - CAIMED Center - Ponce School of Medicine ( Site 0053), Ponce
  - San Juan Hospital ( Site 0056), San Juan
  - University of Puerto Rico ( Site 0051), San Juan
- Thailand (4):
  - Srinagarind Hospital. Khon Kaen University ( Site 0093), Muang, Changwat Khon Kaen
  - Chulalongkorn University ( Site 0092), Bangkok
  - Siriaj Hospital ( Site 0091), Bangkok
  - Maharaj Nakorn Chiang Mai Hospital ( Site 0090), Chiang Mai
- Turkey (Türkiye) (3):
  - Hacettepe University Faculty of Medicine ( Site 0070), Ankara
  - Eskisehir Osmangazi University Faculty of Medicine ( Site 0071), Eskişehir
  - Ege University Medical Faculty Hospital ( Site 0072), Izmir

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bili A, Dobson S, Quinones J, Phongsamart W, Oberdorfer P, Kosalaraksa P, Dagan R, Richmond P, Wilck M, Vallejos W, Nunn C, McFetridge R, Tamms G, Fu R, Lupinacci R, Musey L, Banniettis N, Bickham K; V114-027 PNEU-DIRECTION study group. A phase 3, multicenter, randomized, double-blind study to evaluate the interchangeability of V114, a 15-valent pneumococcal conjugate vaccine, and PCV13 with respect to safety, tolerability, and immunogenicity in healthy infants (PNEU-DIRECTION). Vaccine. 2023 Jan 16;41(3):657-665. doi: 10.1016/j.vaccine.2022.10.072. Epub 2022 Dec 13. PMID 36522265

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were screened at Study Day 1, prior to randomization.
Groups:
- Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™: Participants received a single 0.5 mL intramuscular (IM) injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants concomitantly received other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
- Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and a single 0.5 mL IM injection of V114 on Months 10-13 (Vaccination 4). Participants concomitantly received other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
- Group 3: Prevnar 13™-Prevnar 13™-V114-V114: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2) and a single 0.5 mL IM injection of V114 on Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants concomitantly received other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
- Group 4: Prevnar 13™-V114-V114-V114: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of V114 on Month 2 (Vaccination 2), Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants concomitantly received other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
- Group 5: V114-V114-V114-V114: Participants received a single 0.5 mL IM injection of V114 on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants concomitantly received other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
Period: Overall Study
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Started | 179 | 181 | 180 | 180 | 180
Vaccination 1 (V114 or Prevnar 13™) | 179 | 181 | 178 | 179 | 179
Vaccination 2 (V114 or Prevnar 13™) | 176 | 175 | 166 | 169 | 173
Vaccination 3 (V114 or Prevnar 13™) | 175 | 174 | 161 | 167 | 173
Vaccination 4 (V114 or Prevnar 13™) | 165 | 168 | 150 | 162 | 168
Completed | 164 | 167 | 147 | 160 | 167
Not Completed | 15 | 14 | 33 | 20 | 13
Not completed — Physician Decision | 4 | 0 | 1 | 0 | 2
Not completed — Lost to Follow-up | 2 | 6 | 7 | 3 | 2
Not completed — Consent withdrawn by parent/guardian | 9 | 8 | 25 | 17 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114 | Total
Number analyzed (Participants) | 179 | 181 | 180 | 180 | 180 | 900
Age, Continuous [Mean (Standard Deviation); unit: days] | 63.0 (7.8) | 63.6 (8.4) | 62.7 (9.1) | 63.4 (9.3) | 64.0 (9.3) | 63.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 91 | 85 | 86 | 88 | 426
  Male | 103 | 90 | 95 | 94 | 92 | 474
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 47 | 47 | 43 | 43 | 213
  Not Hispanic or Latino | 146 | 134 | 133 | 136 | 137 | 686
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 36 | 34 | 37 | 32 | 38 | 177
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 | 2
  Black or African American | 8 | 11 | 3 | 3 | 9 | 34
  White | 115 | 106 | 114 | 114 | 104 | 553
  More than one race | 19 | 30 | 26 | 30 | 28 | 133
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Per protocol, the percentage of participants with solicited injection-site AEs was assessed for up to ~14 days after each vaccination. The solicited injection-site AEs assessed were erythema/redness, induration/hard lump, tenderness/pain and swelling.
Time Frame: Up to ~14 days after each vaccination
Population: All randomized participants who got ≥1 dose of V114 or Prevnar 13™.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Number analyzed (Participants) | 179 | 181 | 178 | 179 | 179
Percentage of Participants
  Erythema/Redness | 47.5 | 37.6 | 38.8 | 43.0 | 44.1
  Induration/Hard lump | 34.6 | 26.0 | 28.1 | 25.1 | 26.3
  Tenderness/Pain | 44.1 | 43.6 | 46.1 | 43.6 | 47.5
  Swelling | 22.9 | 18.8 | 24.7 | 20.7 | 22.9
Statistical Analysis 1: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage: Erythema(Group 5 vs 1); Test type: Other — Estimated differences, confidence intervals (CIs), and p-values are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; p = 0.525, Miettinen & Nurminen method; Difference in Percentage = -3.4, 95% CI 2-sided [-13.6 to 7.0]
Statistical Analysis 2: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage: Erythema(Group 4 vs 1); Test type: Other — Estimated differences, CIs, and p-values are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; p = 0.396, Miettinen & Nurminen method; Difference in Percentage = -4.5, 95% CI 2-sided [-14.7 to 5.8]
Statistical Analysis 3: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage: Erythema(Group 3 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.097, Miettinen & Nurminen method; Difference in Percentage = -8.7, 95% CI 2-sided [-18.8 to 1.6]
Statistical Analysis 4: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage: Erythema(Group 2 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.057, Miettinen & Nurminen method; Difference in Percentage = -9.9, 95% CI 2-sided [-19.9 to 0.3]
Statistical Analysis 5: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage: Induration(Group 5 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.085, Miettinen & Nurminen method; Difference in Percentage = -8.4, 95% CI 2-sided [-17.8 to 1.2]
Statistical Analysis 6: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage: Induration(Group 4 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.050, Miettinen & Nurminen method; Difference in Percentage = -9.5, 95% CI 2-sided [-18.9 to -0.0]
Statistical Analysis 7: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage: Induration(Group 3 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.183, Miettinen & Nurminen method; Difference in Percentage = -6.5, 95% CI 2-sided [-16.1 to 3.1]
Statistical Analysis 8: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage: Induration(Group 2 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.074, Miettinen & Nurminen method; Difference in Percentage = -8.7, 95% CI 2-sided [-18.1 to 0.8]
Statistical Analysis 9: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage: Tenderness(Group 5 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.525, Miettinen & Nurminen method; Difference in Percentage = 3.4, 95% CI 2-sided [-7.0 to 13.6]
Statistical Analysis 10: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage: Tenderness(Group 4 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.915, Miettinen & Nurminen method; Difference in Percentage = -0.6, 95% CI 2-sided [-10.8 to 9.7]
Statistical Analysis 11: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage: Tenderness(Group 3 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.714, Miettinen & Nurminen method; Difference in Percentage = 1.9, 95% CI 2-sided [-8.4 to 12.2]
Statistical Analysis 12: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage: Tenderness(Group 2 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.926, Miettinen & Nurminen method; Difference in Percentage = -0.5, 95% CI 2-sided [-10.7 to 9.7]
Statistical Analysis 13: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage: Swelling(Group 5 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p > 0.999, Miettinen & Nurminen method; Difference in Percentage = 0.0, 95% CI 2-sided [-8.7 to 8.7]
Statistical Analysis 14: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage: Swelling(Group 4 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.609, Miettinen & Nurminen method; Difference in Percentage = -2.2, 95% CI 2-sided [-10.8 to 6.4]
Statistical Analysis 15: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage: Swelling(Group 3 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.688, Miettinen & Nurminen method; Difference in Percentage = 1.8, 95% CI 2-sided [-7.1 to 10.7]
Statistical Analysis 16: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage: Swelling(Group 2 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.336, Miettinen & Nurminen method; Difference in Percentage = -4.1, 95% CI 2-sided [-12.6 to 4.3]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Per protocol, the percentage of participants with solicited systemic AEs was assessed for up to ~14 days after each vaccination. The solicited systemic AEs assessed were appetite lost/decreased appetite, irritability, drowsiness/somnolence and hives or welts/urticaria.
Time Frame: Up to ~14 days after each vaccination
Population: All randomized participants who got ≥1 dose of V114 or Prevnar 13™.
Measure: Number; unit: Percentage of Participants
Groups:
- Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and Months 10-13 (Vaccination 4). Participants concomitantly received other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Number analyzed (Participants) | 179 | 181 | 178 | 179 | 179
Percentage of Participants
  Appetite lost/Decreased Appetite | 35.8 | 32.0 | 27.0 | 35.2 | 34.6
  Irritability | 67.6 | 60.8 | 62.9 | 68.2 | 70.4
  Drowsiness/Somnolence | 57.0 | 55.8 | 56.7 | 57.0 | 60.3
  Hives/Urticaria | 7.3 | 3.9 | 5.6 | 8.9 | 6.7
Statistical Analysis 1: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage:Appetite lost(Group5 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.825, Miettinen & Nurminen method; Difference in Percentage = -1.1, 95% CI 2-sided [-11.0 to 8.8]
Statistical Analysis 2: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage:Appetite lost(Group4 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.912, Miettinen & Nurminen method; Difference in Percentage = -0.6, 95% CI 2-sided [-10.4 to 9.3]
Statistical Analysis 3: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage:Appetite lost(Group3 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.074, Miettinen & Nurminen method; Difference in Percentage = -8.8, 95% CI 2-sided [-18.3 to 0.9]
Statistical Analysis 4: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage:Appetite lost(Group2 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.458, Miettinen & Nurminen method; Percentage of Participants = -3.7, 95% CI 2-sided [-13.4 to 6.1]
Statistical Analysis 5: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage:Irritability(Group 5 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.568, Miettinen & Nurminen method; Difference in Percentage = 2.8, 95% CI 2-sided [-6.8 to 12.3]
Statistical Analysis 6: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage:Irritability(Group 4 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.910, Miettinen & Nurminen method; Difference in Percentage = 0.6, 95% CI 2-sided [-9.1 to 10.2]
Statistical Analysis 7: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage:Irritability(Group 3 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.354, Miettinen & Nurminen method; Difference in Percentage = -4.7, 95% CI 2-sided [-14.5 to 5.2]
Statistical Analysis 8: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage:Irritability(Group 2 vs1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.178, Miettinen & Nurminen method; Difference in Percentage = -6.8, 95% CI 2-sided [-16.6 to 3.1]
Statistical Analysis 9: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage: Drowsiness(Group 5 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.520, Miettinen & Nurminen method; Difference in Percentage = 3.4, 95% CI 2-sided [-6.8 to 13.5]
Statistical Analysis 10: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage: Drowsiness(Group 4 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p > 0.999, Miettinen & Nurminen method; Difference in Percentage = 0.0, 95% CI 2-sided [-10.2 to 10.2]
Statistical Analysis 11: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage: Drowsiness(Group 3 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.963, Miettinen & Nurminen method; Difference in Percentage = -0.2, 95% CI 2-sided [-10.5 to 10.0]
Statistical Analysis 12: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage: Drowsiness(Group 2 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.821, Miettinen & Nurminen method; Difference in Percentage = -1.2, 95% CI 2-sided [-11.4 to 9.0]
Statistical Analysis 13: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage: Hives(Group 5 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.836, Miettinen & Nurminen method; Difference in Percentage = -0.6, 95% CI 2-sided [-6.1 to 5.0]
Statistical Analysis 14: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage: Hives(Group 4 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.562, Miettinen & Nurminen method; Difference in Percentage = 1.7, 95% CI 2-sided [-4.2 to 7.6]
Statistical Analysis 15: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage: Hives(Group 3 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.527, Miettinen & Nurminen method; Difference in Percentage = -1.6, 95% CI 2-sided [-7.1 to 3.7]
Statistical Analysis 16: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage: Hives(Group 2 vs 1); Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.160, Miettinen & Nurminen method; Difference in Percentage = -3.4, 95% CI 2-sided [-8.6 to 1.5]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event (SAE)
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires or prolongs existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgement. Relatedness of an SAE to the study vaccine was determined by the investigator. Per protocol, the percentage of participants with vaccine-related SAEs was assessed through 6 months following Vaccination 4.
Time Frame: Up to ~6 months after Vaccination 4 (up to ~19 months)
Population: All randomized participants who got ≥1 dose of V114 or Prevnar 13™.
Measure: Number; unit: Percentage of Participants
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Number analyzed (Participants) | 179 | 181 | 178 | 179 | 179
Percentage of Participants | 0 | 0 | 0.6 | 0 | 0
Statistical Analysis 1: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; Difference in Percentage (Group 5 vs 1); Test type: Other — Estimated differences and CIs are calculated based on the Miettinen & Nurminen method and are provided in accordance with the statistical analysis plan; Difference in Percentage = 0.0, 95% CI 2-sided [-2.1 to 2.1]
Statistical Analysis 2: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; Difference in Percentage (Group 4 vs 1); Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage = 0.0, 95% CI 2-sided [-2.1 to 2.1]
Statistical Analysis 3: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; Difference in Percentage (Group 3 vs 1); Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage = 0.6, 95% CI 2-sided [-1.6 to 3.1]
Statistical Analysis 4: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; Difference in Percentage (Group 2 vs 1); Test type: Other — [test comment as in outcome 3, analysis 1]; Difference in Percentage = 0.0, 95% CI 2-sided [-2.1 to 2.1]

4. Primary Outcome: Geometric Mean Concentration (GMC) of Anti-Pneumococcal Polysaccharide (PnP) Immunoglobulin G (IgG) For 13 Shared Serotypes Contained in V114 and Prevnar 13™ at 30 Days Post Vaccination 4
Description: The GMC of anti-PnP serotype-specific IgG for 13 shared serotypes contained in V114 and Prevnar 13™ (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) was assessed using a pneumococcal electrochemiluminescence (PnECL) assay. Per protocol, 13 IgG serotypes in Groups 2, 3, 4 (experimental arms) were compared to Group 1 (comparator arm) at 30 days post Vaccination 4 as a pre-specified primary outcome analysis; 13 IgG serotypes in Group 5 (experimental arm) were compared to Group 1 (comparator arm) at 30 days post Vaccination 4, as a separate protocol-specified secondary outcome analysis and reported later in the record.
Time Frame: 30 Days after Vaccination 4 (Months 11-14)
Population: All randomized participants who were compliant with the protocol, got scheduled dosing of V114 or Prevnar 13™ and had IgG GMC data for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F or 23F in Groups 1, 2, 3, 4 or 5 at 30 Days post Vaccination 4. 13 IgG serotypes in Groups 2, 3, 4 were compared to Group 1 as a protocol-specified primary outcome analysis; 13 IgG serotypes in Group 5 were compared to Group 1 as a separate protocol-specified secondary outcome analysis and reported later.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Number analyzed (Participants) | 179 | 181 | 178 | 179 | 179
µg/mL
  Serotype 1: number analyzed (Participants) | 147 | 151 | 128 | 139 | 147
  Serotype 1 | 2.02 [1.78 to 2.30] | 1.69 [1.48 to 1.93] | 1.89 [1.63 to 2.18] | 1.68 [1.48 to 1.91] | 1.46 [1.30 to 1.63]
  Serotype 3: number analyzed (Participants) | 148 | 151 | 128 | 139 | 147
  Serotype 3 | 0.72 [0.64 to 0.82] | 0.77 [0.68 to 0.87] | 0.68 [0.61 to 0.77] | 0.73 [0.66 to 0.82] | 0.89 [0.79 to 0.99]
  Serotype 4: number analyzed (Participants) | 146 | 151 | 128 | 139 | 147
  Serotype 4 | 1.51 [1.30 to 1.76] | 1.33 [1.14 to 1.56] | 1.27 [1.10 to 1.46] | 1.23 [1.08 to 1.41] | 1.35 [1.17 to 1.57]
  Serotype 5: number analyzed (Participants) | 147 | 151 | 128 | 138 | 147
  Serotype 5 | 3.66 [3.18 to 4.20] | 3.39 [2.91 to 3.94] | 3.82 [3.23 to 4.51] | 2.90 [2.50 to 3.38] | 2.90 [2.50 to 3.35]
  Serotype 6A: number analyzed (Participants) | 146 | 151 | 128 | 139 | 147
  Serotype 6A | 6.42 [5.56 to 7.42] | 7.16 [6.30 to 8.15] | 7.16 [6.17 to 8.30] | 5.17 [4.43 to 6.03] | 4.43 [3.86 to 5.09]
  Serotype 6B: number analyzed (Participants) | 146 | 151 | 128 | 139 | 147
  Serotype 6B | 6.15 [5.36 to 7.07] | 7.58 [6.61 to 8.68] | 6.64 [5.73 to 7.69] | 6.62 [5.75 to 7.62] | 5.83 [5.09 to 6.68]
  Serotype 7F: number analyzed (Participants) | 146 | 151 | 128 | 139 | 147
  Serotype 7F | 5.10 [4.43 to 5.88] | 5.69 [4.93 to 6.56] | 5.06 [4.33 to 5.92] | 3.98 [3.47 to 4.57] | 3.43 [3.02 to 3.91]
  Serotype 9V: number analyzed (Participants) | 147 | 151 | 128 | 139 | 147
  Serotype 9V | 2.93 [2.56 to 3.34] | 2.76 [2.41 to 3.16] | 2.57 [2.22 to 2.97] | 2.46 [2.19 to 2.78] | 2.89 [2.56 to 3.26]
  Serotype 14: number analyzed (Participants) | 146 | 151 | 128 | 139 | 147
  Serotype 14 | 7.62 [6.55 to 8.86] | 10.59 [9.01 to 12.44] | 10.91 [9.29 to 12.81] | 7.87 [6.77 to 9.16] | 6.57 [5.73 to 7.55]
  Serotype 18C: number analyzed (Participants) | 147 | 151 | 128 | 139 | 147
  Serotype 18C | 2.57 [2.21 to 2.99] | 3.88 [3.38 to 4.45] | 3.70 [3.20 to 4.29] | 2.76 [2.42 to 3.15] | 2.65 [2.34 to 3.01]
  Serotype 19A: number analyzed (Participants) | 148 | 151 | 128 | 139 | 147
  Serotype 19A | 5.92 [5.15 to 6.80] | 5.52 [4.88 to 6.25] | 5.20 [4.42 to 6.12] | 4.95 [4.27 to 5.73] | 4.66 [4.15 to 5.24]
  Serotype 19F: number analyzed (Participants) | 148 | 151 | 128 | 139 | 147
  Serotype 19F | 4.78 [4.22 to 5.42] | 4.88 [4.33 to 5.51] | 5.02 [4.40 to 5.73] | 4.60 [4.00 to 5.28] | 4.10 [3.66 to 4.59]
  Serotype 23F: number analyzed (Participants) | 146 | 150 | 127 | 138 | 146
  Serotype 23F | 2.89 [2.42 to 3.44] | 2.72 [2.33 to 3.18] | 2.29 [1.93 to 2.70] | 2.22 [1.92 to 2.56] | 2.11 [1.81 to 2.46]
Statistical Analysis 1: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 1 (Group 4 vs 1); Test type: Other — GMC ratio and CI are estimated from a serotype-specific ANCOVA model utilizing the natural log-transformed antibody concentration as the response and vaccination group and stratification factor as covariates; GMC Ratio = 0.83, 95% CI 2-sided [0.69 to 1.00]
Statistical Analysis 2: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 1 (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.93, 95% CI 2-sided [0.77 to 1.12]
Statistical Analysis 3: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 1 (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.83, 95% CI 2-sided [0.70 to 1.00]
Statistical Analysis 4: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 3 (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.01, 95% CI 2-sided [0.86 to 1.19]
Statistical Analysis 5: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 3 (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.94, 95% CI 2-sided [0.80 to 1.12]
Statistical Analysis 6: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 3 (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.06, 95% CI 2-sided [0.90 to 1.25]
Statistical Analysis 7: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 4 (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.81, 95% CI 2-sided [0.66 to 1.00]
Statistical Analysis 8: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 4 (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.84, 95% CI 2-sided [0.68 to 1.03]
Statistical Analysis 9: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 4 (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.88, 95% CI 2-sided [0.72 to 1.08]
Statistical Analysis 10: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 5 (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.79, 95% CI 2-sided [0.64 to 0.98]
Statistical Analysis 11: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 5 (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.04, 95% CI 2-sided [0.84 to 1.29]
Statistical Analysis 12: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 5 (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.92, 95% CI 2-sided [0.75 to 1.14]
Statistical Analysis 13: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 6A (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.80, 95% CI 2-sided [0.66 to 0.98]
Statistical Analysis 14: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 6A (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.11, 95% CI 2-sided [0.91 to 1.37]
Statistical Analysis 15: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 6A (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.12, 95% CI 2-sided [0.92 to 1.36]
Statistical Analysis 16: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 6B (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.08, 95% CI 2-sided [0.88 to 1.31]
Statistical Analysis 17: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 6B (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.08, 95% CI 2-sided [0.88 to 1.32]
Statistical Analysis 18: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 6B (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.23, 95% CI 2-sided [1.02 to 1.49]
Statistical Analysis 19: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 7F (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.78, 95% CI 2-sided [0.64 to 0.95]
Statistical Analysis 20: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 7F (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.99, 95% CI 2-sided [0.81 to 1.21]
Statistical Analysis 21: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 7F (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.11, 95% CI 2-sided [0.92 to 1.35]
Statistical Analysis 22: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 9V (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.84, 95% CI 2-sided [0.70 to 1.01]
Statistical Analysis 23: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 9V (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.88, 95% CI 2-sided [0.73 to 1.06]
Statistical Analysis 24: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 9V (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.94, 95% CI 2-sided [0.79 to 1.13]
Statistical Analysis 25: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 14 (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.03, 95% CI 2-sided [0.83 to 1.28]
Statistical Analysis 26: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 14 (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.43, 95% CI 2-sided [1.15 to 1.78]
Statistical Analysis 27: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 14 (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.39, 95% CI 2-sided [1.13 to 1.71]
Statistical Analysis 28: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 18C (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.07, 95% CI 2-sided [0.88 to 1.30]
Statistical Analysis 29: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 18C (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.44, 95% CI 2-sided [1.18 to 1.76]
Statistical Analysis 30: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 18C (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.51, 95% CI 2-sided [1.25 to 1.83]
Statistical Analysis 31: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 19A (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.84, 95% CI 2-sided [0.69 to 1.01]
Statistical Analysis 32: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 19A (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.88, 95% CI 2-sided [0.72 to 1.07]
Statistical Analysis 33: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 19A (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.93, 95% CI 2-sided [0.77 to 1.13]
Statistical Analysis 34: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 19F (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.96, 95% CI 2-sided [0.81 to 1.15]
Statistical Analysis 35: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 19F (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.05, 95% CI 2-sided [0.88 to 1.26]
Statistical Analysis 36: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 19F (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.02, 95% CI 2-sided [0.86 to 1.21]
Statistical Analysis 37: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 4: Prevnar 13™-V114-V114-V114; GMC Ratio: Serotype 23F (Group 4 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.77, 95% CI 2-sided [0.61 to 0.96]
Statistical Analysis 38: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 3: Prevnar 13™-Prevnar 13™-V114-V114; GMC Ratio: Serotype 23F (Group 3 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.79, 95% CI 2-sided [0.63 to 0.99]
Statistical Analysis 39: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114; GMC Ratio: Serotype 23F (Group 2 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.94, 95% CI 2-sided [0.76 to 1.17]

5. Secondary Outcome: Group 5 Versus Group 1 + Group 2: Percentage of Participants With Anti-Hepatitis B Surface Antigen (HBsAg) ≥10 mIU/mL at 30 Days Post Vaccination 3
Description: The concentration of anti-HBsAg was assessed using an enhanced chemiluminescence assay. The protocol-specified analysis of the percentage of participants with anti-HBsAg ≥10 mIU/mL at 30 days post vaccination 3 was conducted in participants combined across vaccine dosing schedules (Group 1 + Group 2) as well as in participants separated across vaccine dosing schedules (Group 1, Group 2). Per protocol, participants with anti-HBsAg ≥10 mIU/mL in Group 5 were compared to Group 1 + Group 2 at 30 days post Vaccination 3, as a pre-specified secondary outcome analysis. Analysis of participants with anti-HBsAg ≥10 mIU/mL was not planned to be reported in Group 3 and Group 4, per protocol.
Time Frame: 30 Days after Vaccination 3 (Month 5)
Population: All randomized participants who were protocol compliant, got scheduled dosing of V114, Prevnar 13™ or background RECOMBIVAX HB™, had anti-HBsAg data at 30 days post Vaccination 3. Per protocol anti-HBsAg analysis was done in participants combined across dosing schedules (Group 1 + 2) and separated across dosing schedules (Group 1, 2). Per protocol Group 5 was compared to Group 1 + 2 as a secondary outcome analysis. Per protocol anti-HBsAg analysis was not planned to be reported in Groups 3, 4.
Measure: Number; unit: Percentage of Participants
Groups:
- Group 1: Prevnar 13™(Vaccinations 1-4) + Group 2: Prevnar 13™(Vaccinations 1-3)-V114 (Vaccination 4): Group 1 participants who received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3), Months 10-13 (Vaccination 4) and Group 2 participants who received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1), Month 2 (Vaccination 2), Month 4 (Vaccination 3) and a single 0.5 mL IM injection of V114 on Months 10-13 (Vaccination 4), were combined across vaccination schedule. Group 1 plus Group 2 participants concomitantly received other licensed background pediatric vaccines as follows: RotaTeq™, Pentacel™, RECOMBIVAX HB™ on Day 1, Month 2, and on Month 4; HIBERIX™, M-M-R™ II, VARIVAX™ on Months 10-13.
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114 | Group 1: Prevnar 13™(Vaccinations 1-4) + Group 2: Prevnar 13™(Vaccinations 1-3)-V114 (Vaccination 4)
Number analyzed (Participants) | 142 | 142 | 0 | 0 | 153 | 284
Percentage of Participants | 98.6 | 99.3 |  |  | 98.7 | 98.9
Statistical Analysis 1: Comparison: Group 5: V114-V114-V114-V114 vs Group 1: Prevnar 13™(Vaccinations 1-4) + Group 2: Prevnar 13™(Vaccinations 1-3)-V114 (Vaccination 4); Difference in Percentage (Group 5 vs Group 1+2); Test type: Non-Inferiority — The statistical criterion for non-inferiority requires the lower bound of the 2-sided 95% CI for the difference in percentages (Group 5/Group 1+Group 2) to be >-10 percentage points; p < 0.001, Miettinen & Nurminen method; Difference in Percentage = -0.2, 95% CI 2-sided [-3.7 to 2.0]

6. Secondary Outcome: Group 5 Versus Group 1 + Group 2: Geometric Mean Titer (GMT) of Anti-Rotavirus Immunoglobulin A (IgA) at 30 Days Post Vaccination 3
Description: The GMT of anti-rotavirus IgA was assessed using a serum IgA enzyme linked immunosorbent assay. The protocol specified analysis of anti-rotavirus IgA GMT at 30 days post vaccination 3 was conducted in participants combined across vaccine dosing schedules (Group 1 + Group 2) as well as in participants separated across vaccine dosing schedules (Group 1, Group 2). Per protocol, GMT of anti-rotavirus IgA in Group 5 was compared to Group 1 + Group 2 at 30 days post Vaccination 3, as a pre-specified secondary outcome analysis. Anti-rotavirus IgA GMT analysis was not planned to be reported in Group 3 and Group 4, per protocol.
Time Frame: 30 Days after Vaccination 3 (Month 5)
Population: All randomized participants who were protocol compliant, got scheduled dosing of V114, Prevnar 13™ or background RotaTeq™, had anti-rotavirus data at 30 days post Vaccination 3. Per protocol anti-rotavirus analysis was done in participants combined across dosing schedules (Group 1 + 2) and separated across dosing schedules (Group 1, 2). Per protocol Group 5 was compared to Group 1 + 2 as a secondary outcome analysis. Per protocol anti-rotavirus analysis was not planned or reported in Group 3, 4
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114 | Group 1: Prevnar 13™(Vaccinations 1-4) + Group 2: Prevnar 13™(Vaccinations 1-3)-V114 (Vaccination 4)
Number analyzed (Participants) | 147 | 143 | 0 | 0 | 152 | 290
Titers | 286.5 [218.1 to 376.2] | 329.5 [254.9 to 426.1] |  |  | 298.3 [228.2 to 390.0] | 307.0 [254.7 to 369.9]
Statistical Analysis 1: Comparison: Group 5: V114-V114-V114-V114 vs Group 1: Prevnar 13™(Vaccinations 1-4) + Group 2: Prevnar 13™(Vaccinations 1-3)-V114 (Vaccination 4); GMT Ratio (Group 5 vs Group 1+2); Test type: Non-Inferiority — The statistical criterion for non-inferiority requires the lower bound of the 2-sided 95% CI for the GMT ratio (Group 5/Group 1+Group 2) to be >0.5; p < 0.001, ANCOVA; GMT Ratio = 0.97, 95% CI 2-sided [0.70 to 1.34]

7. Secondary Outcome: GMC of Anti-PnP IgG for 15 Serotypes Contained in V114 at 30 Days Post Vaccination 3
Description: The concentration of anti-PnP serotype-specific IgG for 15 serotypes contained in V114 (13 serotypes shared with Prevnar 13™ [1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F] and 2 unique serotypes [22F, 33F]) was assessed using a PnECL assay. Per protocol, GMC of 15 IgG serotypes was assessed at 30 days post Vaccination 3.
Time Frame: 30 Days after Vaccination 3 (Month 5)
Population: All randomized participants who were compliant with the protocol, got scheduled dosing of V114 or Prevnar 13™, had IgG GMC data available for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 22F or 33F in Groups 1, 2, 3, 4 or 5 at 30 Days post Vaccination 3.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Number analyzed (Participants) | 179 | 181 | 178 | 179 | 179
µg/mL
  Serotype 1: number analyzed (Participants) | 142 | 142 | 129 | 138 | 148
  Serotype 1 | 1.93 [1.69 to 2.20] | 1.99 [1.78 to 2.21] | 1.86 [1.64 to 2.10] | 1.35 [1.19 to 1.53] | 1.27 [1.14 to 1.41]
  Serotype 3: number analyzed (Participants) | 142 | 142 | 129 | 138 | 147
  Serotype 3 | 0.54 [0.47 to 0.61] | 0.64 [0.56 to 0.73] | 0.56 [0.49 to 0.63] | 0.67 [0.60 to 0.76] | 1.01 [0.91 to 1.12]
  Serotype 4: number analyzed (Participants) | 141 | 139 | 128 | 137 | 147
  Serotype 4 | 1.39 [1.22 to 1.57] | 1.47 [1.30 to 1.66] | 1.34 [1.14 to 1.56] | 1.07 [0.93 to 1.22] | 1.40 [1.24 to 1.57]
  Serotype 5: number analyzed (Participants) | 141 | 141 | 128 | 138 | 148
  Serotype 5 | 1.99 [1.69 to 2.34] | 2.16 [1.87 to 2.49] | 2.15 [1.83 to 2.52] | 1.73 [1.50 to 1.99] | 1.91 [1.67 to 2.18]
  Serotype 6A: number analyzed (Participants) | 140 | 140 | 128 | 138 | 148
  Serotype 6A | 3.07 [2.66 to 3.54] | 3.22 [2.83 to 3.67] | 3.26 [2.79 to 3.82] | 2.05 [1.76 to 2.38] | 1.82 [1.59 to 2.09]
  Serotype 6B: number analyzed (Participants) | 138 | 140 | 127 | 138 | 147
  Serotype 6B | 2.03 [1.66 to 2.49] | 2.50 [2.10 to 2.99] | 2.43 [2.05 to 2.88] | 2.29 [1.91 to 2.76] | 2.26 [1.87 to 2.73]
  Serotype 7F: number analyzed (Participants) | 142 | 142 | 129 | 138 | 148
  Serotype 7F | 3.36 [2.99 to 3.77] | 3.54 [3.16 to 3.96] | 3.52 [3.10 to 3.99] | 2.61 [2.33 to 2.94] | 2.41 [2.17 to 2.67]
  Serotype 9V: number analyzed (Participants) | 143 | 142 | 128 | 138 | 148
  Serotype 9V | 1.69 [1.48 to 1.94] | 1.81 [1.60 to 2.05] | 1.68 [1.44 to 1.97] | 1.47 [1.28 to 1.67] | 2.01 [1.80 to 2.24]
  Serotype 14: number analyzed (Participants) | 142 | 142 | 128 | 138 | 148
  Serotype 14 | 6.57 [5.55 to 7.79] | 6.18 [5.22 to 7.31] | 9.32 [7.45 to 11.67] | 6.71 [5.76 to 7.83] | 5.50 [4.79 to 6.31]
  Serotype 18C: number analyzed (Participants) | 142 | 142 | 129 | 138 | 148
  Serotype 18C | 1.69 [1.46 to 1.95] | 2.03 [1.81 to 2.28] | 2.08 [1.81 to 2.38] | 1.50 [1.33 to 1.71] | 1.51 [1.34 to 1.72]
  Serotype 19A: number analyzed (Participants) | 143 | 142 | 129 | 138 | 148
  Serotype 19A | 2.17 [1.92 to 2.47] | 2.46 [2.21 to 2.74] | 2.25 [1.95 to 2.60] | 1.64 [1.43 to 1.87] | 1.63 [1.47 to 1.82]
  Serotype 19F: number analyzed (Participants) | 143 | 142 | 128 | 138 | 148
  Serotype 19F | 2.83 [2.51 to 3.18] | 2.90 [2.61 to 3.23] | 3.08 [2.72 to 3.48] | 2.32 [2.06 to 2.62] | 2.21 [2.00 to 2.46]
  Serotype 23F: number analyzed (Participants) | 140 | 140 | 128 | 135 | 147
  Serotype 23F | 1.32 [1.09 to 1.59] | 1.72 [1.49 to 1.99] | 1.22 [1.02 to 1.45] | 1.33 [1.14 to 1.57] | 1.46 [1.25 to 1.69]
  Serotype 22F: number analyzed (Participants) | 138 | 140 | 128 | 137 | 148
  Serotype 22F | 0.05 [0.04 to 0.05] | 0.05 [0.04 to 0.06] | 3.63 [2.91 to 4.52] | 5.94 [5.13 to 6.88] | 5.15 [4.52 to 5.87]
  Serotype 33F: number analyzed (Participants) | 141 | 139 | 127 | 137 | 148
  Serotype 33F | 0.05 [0.05 to 0.06] | 0.05 [0.05 to 0.06] | 0.28 [0.21 to 0.36] | 0.89 [0.70 to 1.14] | 2.22 [1.86 to 2.66]

8. Secondary Outcome: Percentage of Participants With Anti-PnP IgG Concentration ≥0.35 µg/mL for 15 Serotypes Contained in V114 at 30 Days Post Vaccination 3
Description: The concentration of anti-PnP serotype-specific IgG for 15 serotypes contained in V114 (13 serotypes shared with Prevnar 13™ [1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F] and 2 unique serotypes [22F, 33F]) was assessed using a PnECL assay. Per protocol, percentage of participants with anti-PnP IgG concentrations ≥0.35 µg/mL was assessed at 30 days post Vaccination 3.
Time Frame: 30 Days after Vaccination 3 (Month 5)
Population: All randomized participants who were compliant with the protocol, got scheduled dosing of V114 or Prevnar 13™, had IgG concentration ≥0.35µg/mL data available for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F, 22F or 33F in Groups 1, 2, 3, 4 or 5 at 30 Days post Vaccination 3.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Number analyzed (Participants) | 179 | 181 | 178 | 179 | 179
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 142 | 142 | 129 | 138 | 148
  Serotype 1 | 97.9 [94.0 to 99.6] | 100 [97.4 to 100.0] | 99.2 [95.8 to 100.0] | 97.8 [93.8 to 99.5] | 96.6 [92.3 to 98.9]
  Serotype 3: number analyzed (Participants) | 142 | 142 | 129 | 138 | 147
  Serotype 3 | 73.2 [65.2 to 80.3] | 73.9 [65.9 to 80.9] | 79.1 [71.0 to 85.7] | 81.9 [74.4 to 87.9] | 93.9 [88.7 to 97.2]
  Serotype 4: number analyzed (Participants) | 141 | 139 | 128 | 137 | 147
  Serotype 4 | 97.9 [93.9 to 99.6] | 98.6 [94.9 to 99.8] | 93.0 [87.1 to 96.7] | 94.2 [88.8 to 97.4] | 96.6 [92.2 to 98.9]
  Serotype 5: number analyzed (Participants) | 141 | 141 | 128 | 138 | 148
  Serotype 5 | 97.9 [93.9 to 99.6] | 99.3 [96.1 to 100.0] | 97.7 [93.3 to 99.5] | 97.1 [92.7 to 99.2] | 98.0 [94.2 to 99.6]
  Serotype 6A: number analyzed (Participants) | 140 | 140 | 128 | 138 | 148
  Serotype 6A | 99.3 [96.1 to 100.0] | 99.3 [96.1 to 100.0] | 99.2 [95.7 to 100.0] | 97.1 [92.7 to 99.2] | 98.6 [95.2 to 99.8]
  Serotype 6B: number analyzed (Participants) | 138 | 140 | 127 | 138 | 147
  Serotype 6B | 91.3 [85.3 to 95.4] | 94.3 [89.1 to 97.5] | 96.1 [91.1 to 98.7] | 95.7 [90.8 to 98.4] | 95.2 [90.4 to 98.1]
  Serotype 7F: number analyzed (Participants) | 142 | 142 | 129 | 138 | 148
  Serotype 7F | 100 [97.4 to 100.0] | 100 [97.4 to 100] | 100 [97.2 to 100.0] | 100 [97.4 to 100.0] | 100 [97.5 to 100.0]
  Serotype 9V: number analyzed (Participants) | 143 | 142 | 128 | 138 | 148
  Serotype 9V | 96.5 [92.0 to 98.9] | 96.5 [92.0 to 98.8] | 96.1 [91.1 to 98.7] | 95.7 [90.8 to 98.4] | 98.6 [95.2 to 99.8]
  Serotype 14: number analyzed (Participants) | 142 | 142 | 128 | 138 | 148
  Serotype 14 | 98.6 [95.0 to 99.8] | 98.6 [95.0 to 99.8] | 96.9 [92.2 to 99.1] | 100 [97.4 to 100.0] | 98.6 [95.2 to 99.8]
  Serotype 18C: number analyzed (Participants) | 142 | 142 | 129 | 138 | 148
  Serotype 18C | 95.8 [91.0 to 98.4] | 100 [97.4 to 100.0] | 99.2 [95.8 to 100.0] | 97.8 [93.8 to 99.5] | 98.0 [94.2 to 99.6]
  Serotype 19A: number analyzed (Participants) | 143 | 142 | 129 | 138 | 148
  Serotype 19A | 99.3 [96.2 to 100.0] | 100 [97.4 to 100.0] | 98.4 [94.5 to 99.8] | 97.1 [92.7 to 99.2] | 97.3 [93.2 to 99.3]
  Serotype 19F: number analyzed (Participants) | 143 | 142 | 128 | 138 | 148
  Serotype 19F | 99.3 [96.2 to 100.0] | 99.3 [96.1 to 100.0] | 99.2 [95.7 to 100.0] | 100 [97.4 to 100.0] | 100 [97.5 to 100.0]
  Serotype 23F: number analyzed (Participants) | 140 | 140 | 128 | 135 | 147
  Serotype 23F | 91.4 [85.5 to 95.5] | 97.9 [93.9 to 99.6] | 90.6 [84.2 to 95.1] | 92.6 [86.8 to 96.4] | 94.6 [89.6 to 97.6]
  Serotype 22F: number analyzed (Participants) | 138 | 140 | 128 | 137 | 148
  Serotype 22F | 2.9 [0.8 to 7.3] | 1.4 [0.2 to 5.1] | 93.8 [88.1 to 97.3] | 99.3 [96.0 to 100.0] | 98.6 [95.2 to 99.8]
  Serotype 33F: number analyzed (Participants) | 141 | 139 | 127 | 137 | 148
  Serotype 33F | 2.1 [0.4 to 6.1] | 2.2 [0.4 to 6.2] | 39.4 [30.8 to 48.4] | 75.9 [67.9 to 82.8] | 93.2 [87.9 to 96.7]

9. Secondary Outcome: Group 5 Versus Group 1: GMC of Anti-PnP IgG For 13 Shared Serotypes Contained in V114 and Prevnar 13™ at 30 Days Post Vaccination 4
Description: The GMC of anti-PnP serotype-specific IgG for 13 shared serotypes contained in V114 and Prevnar 13™ (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) was assessed using a PnECL assay. Per protocol, GMC of 13 IgG serotypes was analysed by vaccine dosing schedules (Groups 1, 5). Per protocol, 13 IgG serotypes in Group 5 (experimental arm) were compared to Group 1 (comparator arm) at 30 days post Vaccination 4 as a pre-specified secondary outcome analysis; 13 IgG serotypes in Groups 2, 3, 4 (experimental arms) were compared to Group 1 (comparator arm) at 30 days post Vaccination 4, as a separate protocol-specified primary outcome analysis and reported earlier in the record.
Time Frame: 30 Days after Vaccination 4 (Months 11-14)
Population: All randomized participants who were compliant with the protocol, got scheduled dosing of V114 or Prevnar 13™, had IgG GMC data available for serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F or 23F in Groups 5 or 1 at 30 Days post Vaccination 4. 13 IgG serotypes in Group 5 were compared to Group 1 as a protocol-specified secondary outcome analysis; 13 IgG serotypes in Groups 2, 3, 4 were compared to Group 1 as a separate protocol-specified primary outcome analysis and reported earlier.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
Number analyzed (Participants) | 179 | 0 | 0 | 0 | 179
µg/mL
  Serotype 1: number analyzed (Participants) | 147 | 0 | 0 | 0 | 147
  Serotype 1 | 2.02 [1.78 to 2.30] |  |  |  | 1.46 [1.30 to 1.63]
  Serotype 3: number analyzed (Participants) | 148 | 0 | 0 | 0 | 147
  Serotype 3 | 0.72 [0.64 to 0.82] |  |  |  | 0.89 [0.79 to 0.99]
  Serotype 4: number analyzed (Participants) | 146 | 0 | 0 | 0 | 147
  Serotype 4 | 1.51 [1.30 to 1.76] |  |  |  | 1.35 [1.17 to 1.57]
  Serotype 5: number analyzed (Participants) | 147 | 0 | 0 | 0 | 147
  Serotype 5 | 3.66 [3.18 to 4.20] |  |  |  | 2.90 [2.50 to 3.35]
  Serotype 6A: number analyzed (Participants) | 146 | 0 | 0 | 0 | 147
  Serotype 6A | 6.42 [5.56 to 7.42] |  |  |  | 4.43 [3.86 to 5.09]
  Serotype 6B: number analyzed (Participants) | 146 | 0 | 0 | 0 | 147
  Serotype 6B | 6.15 [5.36 to 7.07] |  |  |  | 5.83 [5.09 to 6.68]
  Serotype 7F: number analyzed (Participants) | 146 | 0 | 0 | 0 | 147
  Serotype 7F | 5.10 [4.43 to 5.88] |  |  |  | 3.43 [3.02 to 3.91]
  Serotype 9V: number analyzed (Participants) | 147 | 0 | 0 | 0 | 147
  Serotype 9V | 2.93 [2.56 to 3.34] |  |  |  | 2.89 [2.56 to 3.26]
  Serotype 14: number analyzed (Participants) | 146 | 0 | 0 | 0 | 147
  Serotype 14 | 7.62 [6.55 to 8.86] |  |  |  | 6.57 [5.73 to 7.55]
  Serotype 18C: number analyzed (Participants) | 147 | 0 | 0 | 0 | 147
  Serotype 18C | 2.57 [2.21 to 2.99] |  |  |  | 2.65 [2.34 to 3.01]
  Serotype 19A: number analyzed (Participants) | 148 | 0 | 0 | 0 | 147
  Serotype 19A | 5.92 [5.15 to 6.80] |  |  |  | 4.66 [4.15 to 5.24]
  Serotype 19F: number analyzed (Participants) | 148 | 0 | 0 | 0 | 147
  Serotype 19F | 4.78 [4.22 to 5.42] |  |  |  | 4.10 [3.66 to 4.59]
  Serotype 23F: number analyzed (Participants) | 146 | 0 | 0 | 0 | 146
  Serotype 23F | 2.89 [2.42 to 3.44] |  |  |  | 2.11 [1.81 to 2.46]
Statistical Analysis 1: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 1 (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.72, 95% CI 2-sided [0.60 to 0.86]
Statistical Analysis 2: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 3 (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.22, 95% CI 2-sided [1.04 to 1.44]
Statistical Analysis 3: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 4 (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.89, 95% CI 2-sided [0.73 to 1.10]
Statistical Analysis 4: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 5 (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.79, 95% CI 2-sided [0.64 to 0.97]
Statistical Analysis 5: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 6A (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.69, 95% CI 2-sided [0.57 to 0.84]
Statistical Analysis 6: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 6B (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.95, 95% CI 2-sided [0.78 to 1.15]
Statistical Analysis 7: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 7F (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.67, 95% CI 2-sided [0.55 to 0.82]
Statistical Analysis 8: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 9V (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.99, 95% CI 2-sided [0.82 to 1.18]
Statistical Analysis 9: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 14 (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.86, 95% CI 2-sided [0.70 to 1.07]
Statistical Analysis 10: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 18C (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 1.03, 95% CI 2-sided [0.85 to 1.25]
Statistical Analysis 11: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 19A (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.79, 95% CI 2-sided [0.65 to 0.95]
Statistical Analysis 12: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 19F (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.86, 95% CI 2-sided [0.72 to 1.02]
Statistical Analysis 13: Comparison: Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ vs Group 5: V114-V114-V114-V114; GMC Ratio: Serotype 23F (Group 5 vs 1); Test type: Other — [test comment as in outcome 4, analysis 1]; GMC Ratio = 0.73, 95% CI 2-sided [0.59 to 0.91]

ADVERSE EVENTS:
Time Frame: Non-serious AEs (NSAEs): Up to ~14 days after each vaccination; SAEs and all-cause mortality: Up to ~6 months after Vaccination 4 (up to ~19 months)
Description: All-cause mortality was analyzed in all randomized participants; SAEs and NSAEs were analyzed in all randomized participants who received at least 1 dose of study vaccination V114 or Prevnar 13™.
Arm/Group | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 | Group 4: Prevnar 13™-V114-V114-V114 | Group 5: V114-V114-V114-V114
All-Cause Mortality (participants affected / at risk) | 0/179 | 0/181 | 0/180 | 0/180 | 0/180
Serious Adverse Events (participants affected / at risk) | 21/179 | 24/181 | 15/178 | 18/179 | 21/179
Other Adverse Events (participants affected / at risk) | 164/179 | 161/181 | 160/178 | 163/179 | 160/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ (N=179) | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 (N=181) | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 (N=178) | Group 4: Prevnar 13™-V114-V114-V114 (N=179) | Group 5: V114-V114-V114-V114 (N=179)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenoviral upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 6 (6) | 6 (6) | 3 (3) | 3 (3) | 8 (8)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Exanthema subitum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpangina (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Mycoplasma infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 3 (3)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair follicle tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Prevnar 13™-Prevnar 13™-Prevnar 13™-Prevnar 13™ (N=179) | Group 2: Prevnar 13™-Prevnar 13™-Prevnar 13™-V114 (N=181) | Group 3: Prevnar 13™-Prevnar 13™-V114-V114 (N=178) | Group 4: Prevnar 13™-V114-V114-V114 (N=179) | Group 5: V114-V114-V114-V114 (N=179)
Diarrhoea (Gastrointestinal disorders) | 15 (20) | 11 (12) | 11 (12) | 10 (10) | 10 (12)
Vomiting (Gastrointestinal disorders) | 8 (11) | 11 (12) | 4 (4) | 11 (13) | 11 (11)
Injection site erythema (General disorders) | 85 (137) | 68 (108) | 69 (109) | 77 (130) | 79 (142)
Injection site induration (General disorders) | 62 (106) | 47 (83) | 50 (84) | 45 (75) | 47 (86)
Injection site pain (General disorders) | 79 (158) | 79 (140) | 82 (165) | 78 (156) | 85 (170)
Injection site swelling (General disorders) | 41 (58) | 34 (55) | 44 (63) | 37 (59) | 41 (71)
Pyrexia (General disorders) | 53 (83) | 66 (94) | 52 (77) | 49 (78) | 49 (68)
Nasopharyngitis (Infections and infestations) | 10 (12) | 11 (12) | 13 (14) | 8 (8) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 9 (10) | 9 (11) | 12 (13) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 64 (150) | 58 (95) | 48 (77) | 63 (90) | 62 (121)
Somnolence (Nervous system disorders) | 102 (285) | 101 (241) | 101 (207) | 102 (248) | 108 (237)
Irritability (Psychiatric disorders) | 121 (430) | 110 (362) | 112 (378) | 122 (376) | 126 (434)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 12 (14) | 10 (13) | 18 (20) | 17 (17)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 15 (18) | 12 (14) | 12 (16) | 14 (15)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (4) | 16 (16) | 6 (6)
Urticaria (Skin and subcutaneous tissue disorders) | 13 (16) | 7 (9) | 10 (14) | 16 (20) | 12 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03620162/Prot_SAP_000.pdf